CLINICAL TRIAL: NCT06606249
Title: Randomized Trial of a Brief, Transdiagnostic, Guided Self-help Intervention for University Students Who Are Behind on Their Coursework and Experience Distress
Brief Title: Self-Help Plus for Distress in University Students
Acronym: SSH+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Universita di Verona (Other); University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, CRISTEA IOANA ALINA, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20224XSWRH
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Psychological Distress; Psychological Well-Being; Depression; Anxiety
Keywords: prevention; university students; academic deceit; emotion regulation
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Emotional Regulation | interventions — Psychological First Aid

STUDY DESIGN:
Intervention Model Description: The study will involve three centers (Padova, Verona, Bari). Randomization will be individual and stratified by the three recruiting center, with an allocation rate of 1:1:1. A centralized system (Redcap) will be used to generate the randomization schedule, using randomly permuted blocks of unequal size.
Who Masked: Investigator
Masking Description: The three site investigators will not be made aware of the block size or have any access to the randomization schedule. The software allows for random allocation of participants after the baseline evaluation is performed and inclusion criteria are checked. The study statistician will also be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Help Plus (SH+) (Experimental): The intervention is available in its individual online self-help version called "Doing What Matters in Time of Stress". It composed of an illustrate guide, divided into sessions, and pre-recorded audio.
  Participants will be required to access an online platform for attending the sessions. A total of 5 sessions of approximately an hour each are planned. Participants will be guided by facilitators with minimal qualifications and skills in providing psychosocial support. They will receive regular reminders and instructions from helpers at the beginning of the program and before any sessions via phone call, teleconferencing meeting, or message. Facilitators will receive brief training from specialized mental health professionals trained by WHO.
  Interventions: Behavioral: Self-Help Plus (SH+)
- Psychological First Aid (PFA) (Active Comparator): Psychological First Aid will also be delivered by facilitators through a phone call or teleconferencing meeting, for an approximate ranging from 20 to 45 minutes. Participants will also receive an information sheet with details about mental health services available for students experiencing distress at each of the centers.
  Interventions: Behavioral: Psychological First Aid (PFA)

INTERVENTIONS:
Behavioral: Self-Help Plus (SH+) — Self-Help Plus is a novel, brief, low-intensity intervention, recently developed by the World Health Organization (WHO) and intended to help people with and without mental disorders cope with distress stemming from diverse types of adversity.The key components of the program are based on acceptance and commitment therapy (ACT), a distinct form of cognitive-behavioural therapy. SH+ draws on ACT techniques of coping with stress, compassion and acceptance toward oneself and others, and living following one's values.
  An online version called "Doing what matters in times of stress" is available as an illustrated guide and pre-recorded audio.
  Other Names: Doing what matters in times of stress
  Arms: Self-Help Plus (SH+)
Behavioral: Psychological First Aid (PFA) — Psychological First Aid (PFA) is also developed by the WHO and is a general supportive intervention, aimed at listening and understanding the needs and concerns of people, providing support without pressuring them to talk.
  Arms: Psychological First Aid (PFA)

SUMMARY:
Prrospective, multi-center, randomized controlled trial of a brief, transdiagnostic, guided self-help intervention (Self-Help Plus) for university students who experience significant distress and are behind on their coursework. The intervention will be tested in terms of efficacy and feasibility for outcomes related to distress, anxiety, depression and well-being, assessed immediately after the intervention and at 3-months follow-up.

DETAILED DESCRIPTION:
The university period usually overlaps with a particularly challenging developmental period of transition to adulthood, and a suite of significant and durable stressors, such as independent living, financial problems, interpersonal relationships with family or peers and academic pressure. Consequently, it represents a critical high-risk period for the onset of mental disorders, including anxiety, depression, substance abuse, self-harm and suicidal behavior. In the World Mental Health Surveys, a set of large-scale cross-national community epidemiological surveys, the 12-month prevalence of any mental disorder among university students was around 20%. Further compounding the problem, a large survey on first year university students in high-income countries showed that approximately 36% of students with any lifetime mental disorder or with suicidal thoughts or behaviors had received any treatment for emotional problems in the past year. Lack of awareness of the problem and fear of stigma might account for the low treatment uptake in university students.

Furthermore, university psychological counseling services, when available, have limited impact, due to their isolation from the general health care system and to the heterogeneity of the interventions offered. An alternative, innovative framework to promote access to mental health interventions while minimizing the risk of stigmatization is "indirect prevention". This approach includes interventions that address vulnerability factors increasing the risk of mental disorders while at the same time representing salient, everyday problems that students are motivated to change. In a diathesis-stress model, mental disorders are triggered by the interaction between individual vulnerability factors and stressors such as academic challenges.

A promising candidate intervention is Self-Help Plus (SH+), developed by the World Health Organization (WHO) and intended to help individuals cope with distress stemming from a diversity of stressors. In its individual online version called Doing What Matters in Times of Stress, SH+ might be particularly suitable for university students given its easily implementable structure (5 sessions of guided self-help), its contents (focused on self-compassion, coping with stress and personal values), and delivery format (not requiring specialized training). Only two randomized trials so far employed SH+ as a preventive intervention, targeting refugees in Western Europe and Turkey. This is the first attempt to test SH+ as a preventive intervention on university students.

ELIGIBILITY:
Inclusion Criteria:

* University students across all years of higher education (i.e., bachelor and masters), enrolled in any degree course, starting from the second semester of the 1st year
* Currently behind coursework by at least 3 exams, including: exams failed, for which the obtained grade was not confirmed by the student (i.e., confirming the grade is mandatory in the Italian academic system), or postponed (i.e., not taken in the regularly scheduled period).
* Experience significant distress as assessed by the Kessler psychological distress scale (K-10) ≥ 16.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Kessler psychological distress scale | Baseline, After the intervention, At 3 months after the intervention
  The Kessler psychological distress scale (K-10) is a simple measure of psychological distress. It consists of 10 questions about emotional states that can be answered from 1 (none of the time) to 5 (all of the time). Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline, After the intervention, At 3 months after the intervention
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report instrument to measure depression. It consists of 9 items, each rated on a 4-point scale ranging from 0 (not at all) to 3 (almost every day). Total scores range from 0 to 27.
The Generalized Anxiety Disorder-7 | Baseline, After the intervention, At 3 months after the intervention
  The General Anxiety Disorder-7 (GAD-7) scale is a measure of symptoms of generalized anxiety. It consists of 7 items that can be rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores can range from 0 to 21.
World Health Organization Well-Being Index | Baseline, After the intervention, At 3 months after the intervention
  World Health Organization Well-Being Index (WHO-5) assesses subjective well-being. It consists of 5 items, each rated on a 6-point scale ranging from 0 (at no time) to 5 (all of the time). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, ranging from 0 to 100.
Numbers of exams sustained | Baseline, After the intervention, At 3 months after the intervention
  Self-reported number of exams sustained over the study period
Academic deceit survey | Baseline, After the intervention, At 3 months after the intervention
  An ad hoc tool with three questions will be used: (a) did you lie to significant others about academic status; (b) how frequently, on a scale ranging from 0 (never) to 4 (always) and (c) in which situations (open ended)

OTHER OUTCOMES:
Accesibility | Immediately after the intervention
  Easy access to the online intervention and to the rating scales
Intervention dose | Immediately after the intervention
  Number of sessions attended by each participant, and the time spent in each session measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Cristea, PhD, Principal Investigator — University of Padova
Locations (3):
- Italy (3):
  - University of Bari "Aldo Moro", Bari, Bari
  - University of Padova, Padua
  - Universita di Verona, Verona

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized and de-identified individual participant data will be made available, following a request and the signing of a data sharing agreement, completed by the data requestor and directed to the principal investigator. Complete metadata and analysis scripts will be made publicly available with each publication.
  Individual participant data will be made available for research purposes only, including replication. The data will not be made available for non-research purposes in accordance with the legal framework underpinning ethical approval and informed consent.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year after study completion.
Access Criteria: Interested parties will have to submit a data request including as a minimum the purpose of accessing the data, how the data will be used and how findings will be disseminated. A data sharing agreement will be signed between the requestor and principal investigator underlying the purposes and conditions for which data will be used.